CLINICAL TRIAL: NCT05244824
Title: Adaptation of Evaluation of Daily Activity Questionnaire (EDAQ) Into Turkish, Examining The Reliability and Validity For People With Rheumatoid Arthritis
Brief Title: Adaptation of EDAQ Into Turkish, Examining The Reliability and Validity For People With RA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Collaborators: Büşra Kaplan (Unknown); Alison Hammond (Unknown); Fatma Gün (Unknown); Özgün Belen (Unknown); Remziye Akarsu (Unknown); Gözde Kübra Yardımcı (Unknown); Umut Kalyoncu (Unknown); Mehmet Yusuf Çelik (Unknown)
Responsible Party: Principal Investigator, Gonca Bumin, Prof. Dr., Hacettepe University
Other Study IDs: GO21/203
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Arthritis, Rheumatoid; Activities of Daily Living
Keywords: ADL, RA
MeSH Terms: conditions — Arthritis, Rheumatoid; Sarcoglycanopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis: To translate the EDAQ, which determines the difficulties experienced by individuals with rheumatoid arthritis in daily life, into Turkish.
  Interventions: Other: Adaptation into Turkish, Examining The Reliability and Validity for People with RA

INTERVENTIONS:
Other: Adaptation into Turkish, Examining The Reliability and Validity for People with RA — Adaptation of Evaluation of Daily Activity Questionnaire into Turkish, examining the reliability and validity for people with rheumatoid arthritis

SUMMARY:
The aim of the study is to adapt the Evaluation of Daily Activity Questionnaire into Turkish language, and to examine the reliability and validity for people with rheumatoid arthritis.

DETAILED DESCRIPTION:
Patient-Reported Outcome Measures are used in clinical practice and research to identify patients with rheumatic and musculoskeletal conditions' functional problems and evaluate the effectiveness of rehabilitation for these. Most commonly, daily activities in the International Classification of Functioning, Disability and Health (ICF) domains of communication, mobility, self-care and domestic life are assessed. Measurement tools commonly used in rheumatology out-patient clinics and research (e.g., the Health Assessment Questionnaire and the Arthritis Impact Measurement Scales 2 include too few activities to be of use for treatment planning. The Evaluation of Daily Activity Questionnaire was developed in the early 1990s in Sweden to address these problems. It is a patient-reported outcome measure evaluating common symptoms and measuring, in depth, activity limitations in rheumatoid arthritis. Patients normally complete it at home, allowing them time to reflect on their abilities and activity limitations. It normally takes between 25 and 35 min to complete.

Hammond et al have developed an English Evaluation of Daily Activity Questionnaire, which has been linguistically and culturally validated for use in the UK (from the original Swedish version). This was shown to be psychometrically robust for use with patients with rheumatoid arthritis. Subsequently, Hammond et al established the EDAQ's content validity and acceptability and demonstrated reliability and validity in seven other musculoskeletal conditions: ankylosing spondylitis; osteoarthritis; systemic lupus erythematosus; systemic sclerosis; chronic pain; chronic hand/upper limb musculoskeletal disorders; and primary Sjögren's syndrome. These conditions were selected as more often referred to occupational therapy. An EDAQ User Manual is available.

This questionnaire evaluates daily living activities of patients with arthritis and musculoskeletal conditions very comprehensively. Cross-cultural adaptation of the EDAQ into the Turkish language would enable its use in Turkey to identify the daily living activity problems for patients with rheumatoid arthritis. This questionnaire will be directional in clinical and academic studies.

The aim of the study is to adapt the Evaluation of Daily Activity Questionnaire into Turkish language, and to examine the reliability and validity for people with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age and older
* A confirmed diagnosis of rheumatoid arthritis
* Able to read, write and understand Turkish

Exclusion Criteria:

* Have cognitive impairment affecting ability to understand and complete the study questionnaire.
* Altered their disease-modifying medication regimen in the last 3 months
* Have another neurological or psychiatric diseases that effects daily living activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Since the Rasch analysis was used to evaluate the construct validity, it was determined that regardless of whether the scale was targeted well or not and considering the 99% confidence probability that item estimation was sufficient, a sample size of at least 210 should be taken, and 80 people should be taken for test-retest reliability.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Daily Activities Questionnaire (EDAQ) | 45 minute
  The Evaluation of Daily Activities Questionnaire (EDAQ) was developed to meet the needs of occupational therapists for a valid, reliable and detailed Patient Reported Outcome Measure. It is used in clinical practice in rheumatoid arthritis and other musculoskeletal diseases. It consists of 3 parts. Part 1 includes 10-point numeric rating scales that evaluate the common symptoms and effects of arthritis.Part 2 consists of 14 domains including 138 activities identified by people with rheumatoid arthritis as being often problematic. Twelve of these 14 domains can be combined to form some components: Self-Care, Mobility, Caring and Leisure/social activity. Part 2 corresponds to Activity and Participation in the ICF. Part 3 is optional and includes a checklist of assistive devices.
Health Assessment Questionnaire (HAQ) | 10 minute
  The Health Assessment Questionnaire (HAQ) is an assessment tool created in 1980 to evaluate the daily and physical activities of rheumatoid arthritis patients. It is usually used with rheumatoid arthritis and osteoarthritis patients. The HAQ, which takes about 10 minutes to complete, is completed by the patient. The HAQ contains 20 items classified into eight domains. Items include daily activities such as dressing, eating, sitting up, hygiene, walking, grasping, reaching out. The questionnaire is scored with a 4-point Likert scale: "without any difficulty - 0", "with some difficulty - 1", "with much difficulty - 2", "unable to do - 3". The final score of the HAQ is the total item scores. The minimum possible total score is "0" and the maximum possible total score is "60". A higher score indicates greater disability.
Short Form-36 (SF-36v1) | 15 minute
  Short Form 36v1 is a general health questionnaire that evaluates the perception of quality of life for the last four weeks in eight subcategories and 36 items: Physical functions, physical roles (role limitations because of physical condition), pain, social functions, mental health, emotional roles (role limitations because of emotional condition) energy and perception of general health. Two subgroups have "yes" and "no" answers, the other 6 subgroups use a Likert rating scale. Each subgroup is scored between 0 and 100, with a high score indicating good health. It is a generic measure, that is it can be used to measure and compare outcomes in different diseases and treatments, unlike disease-specific assessments (17). The Turkish SF36v1 has been shown to have good validity and reliability in patients with rheumatoid.
Rheumatoid Arthritis Quality of Life Questionnaire (RAQoL) | 10 minute
  The Rheumatoid Arthritis Quality of Life Questionnaire is a disease-specific scale developed for patients with rheumatoid arthritis and is a multidimensional quality of life scale. It consists of 30 questions answered as yes or no. Scores range from 0 to 30, with a high score indicating low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Bumin, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Demographic and other socio-economic data will be collected and recorded, including age, gender, disease duration, employment status, marital status, living circumstances (alone; with significant others); number and age of children; and current medication.
  Because of the Covid-19 Pandemic and health and safety reasons, the sociodemographic information form, Evaluation of Daily Activity Questionnaire, Health Assessment Questionnaire, SF-36v1 and Rheumatoid Arthritis Quality of Life Questionnaire will be adapted into a Google form questionnaire. The questionnaire will be e-mailed to the participants with rheumatoid arthritis as a Google form questionnaire weblink. For those who do not have access to e-mail and the internet, a paper questionnaire option will be available by mail.

REFERENCES:
- [Result] Hammond A, Tennant A, Tyson SF, Nordenskiold U, Hawkins R, Prior Y. The reliability and validity of the English version of the Evaluation of Daily Activity Questionnaire for people with rheumatoid arthritis. Rheumatology (Oxford). 2015 Sep;54(9):1605-15. doi: 10.1093/rheumatology/kev008. Epub 2015 Apr 10. PMID 25863045
- [Result] Hammond A, Meesters J, Niedermann K, Tennant A, Vliet Vlieland T, Tyson S, Nordenskiold U. Cross-cultural adaptation and psychometric testing of the Dutch and German versions of the Evaluation of Daily Activity Questionnaire in people with rheumatoid arthritis. Rheumatol Int. 2021 May;41(5):951-964. doi: 10.1007/s00296-020-04657-7. Epub 2020 Jul 26. PMID 32715341
- [Result] Hammond A, Tyson S, Prior Y, Hawkins R, Tennant A, Nordenskiold U, Thyberg I, Sandqvist G, Cederlund R. Linguistic validation and cultural adaptation of an English version of the evaluation of daily activity questionnaire in rheumatoid arthritis. Health Qual Life Outcomes. 2014 Sep 20;12:143. doi: 10.1186/s12955-014-0143-y. PMID 25238819
- [Result] Adroher ND, Tennant A. Supporting construct validity of the Evaluation of Daily Activity Questionnaire using Linear Logistic Test Models. Qual Life Res. 2019 Jun;28(6):1627-1639. doi: 10.1007/s11136-019-02146-4. Epub 2019 Mar 9. PMID 30852765
- See also: EDAQ Manual v3 — http://usir.salford.ac.uk/id/eprint/30752/